CLINICAL TRIAL: NCT02256111
Title: EXTEND: Safety and Efficacy of EXercise Training in Men Receiving ENzalutamide in Combination With Conventional Androgen Deprivation Therapy for Hormone Naïve Prostate Cancer
Brief Title: EXTEND Exercise Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053924
Record Dates: First submitted 2014-08-22; First posted 2014-10-03 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-03

CONDITIONS: Non-metastatic, Hormone naïve Prostate Cancer
MeSH Terms: interventions — enzalutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENZ+ADT+Usual care (Experimental): The usual care arm will receive treatment with enzalutamide with androgen deprivation therapy, with no supervised exercise training.
  Interventions: Drug: Enzalutamide; Drug: Androgen deprivation therapy
- ENZ+ADT+Exercise (Experimental): The ENZ+ADT+Exercise arm will receive treatment with enzalutamide plus androgen deprivation therapy along with supervised exercise training.
  Interventions: Drug: Enzalutamide; Drug: Androgen deprivation therapy; Behavioral: Supervised exercise training

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: Xtandi
Drug: Androgen deprivation therapy
Behavioral: Supervised exercise training
  Arms: ENZ+ADT+Exercise

SUMMARY:
This study will examine the effect of supervised exercise training on cardiopulmonary function in men receiving the combination of enzalutamide (ENZ) and androgen deprivation therapy (ADT) for treatment of non-metastatic, hormone-naïve prostate cancer. No study to date has examined the efficacy, tolerability, and safety of exercise training to prevent and/or mitigate common adverse toxicities in men receiving combination androgen suppression therapy for hormone-naïve prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male age ≥ 18 years.
2. Histologically-confirmed adenocarcinoma of the prostate.
3. Completion of appropriate prior treatment with local therapy (i.e., prostatectomy, radiation therapy or equivalent), per NCCN Guidelines.
4. Detectable PSA, defined as PSA ≥0.01 ng/ml
5. Appropriate for treatment with ADT in the opinion of the treating physician.
6. Serum total testosterone ≥150 ng/dL (5.2 nmol/L).
7. ECOG performance status of ≤ 1 (Appendix A)
8. Planned treatment with castration therapy (GnRH agonist/antagonist) for ≥8 months.
9. Must not have any of the following absolute contraindications to cardiopulmonary exercise testing and/or aerobic training as determined by the attending oncologist:

   Absolute Contraindications
   * Acute myocardial Infarction (within 3-5 days of any planned study procedures)
   * Unstable angina
   * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
   * Recurrent syncope
   * Active endocarditis
   * Acute myocarditis or pericarditis
   * Symptomatic severe aortic stenosis
   * Uncontrolled heart failure
   * Acute (within 3 months) pulmonary embolus or pulmonary infarction
   * Thrombosis of lower extremities
   * Suspected dissecting aneurysm
   * Uncontrolled asthma
   * Pulmonary edema
   * Room air desaturation at rest <85%
   * Respiratory failure
   * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e. infection, renal failure, thyrotoxicosis)
   * Mental impairment leading to inability to cooperate.
10. Able to swallow enzalutamide and comply with study requirements.
11. Must be able to complete an acceptable cardiopulmonary exercise test (CPET) at baseline (see Section 9), defined as at least one of the following:

    * Achieving a plateau in oxygen consumption concurrent with an increase in power output;
    * Respiratory exchange ratio ≥ 1.1 (RER);
    * Volitional exhaustion with a rating of perceived exertion ≥ 17 (RPE)
12. Must be able to complete an acceptable muscular strength test (assessed using calculated one-repetition maximum (1-RM)) at baseline (see Section 9), in the opinion of the fitness specialist, exercise physiologist, or trained designee administering the test.
13. Life expectancy of ≥ 12 months.
14. Must use a condom if having sex with a pregnant woman.
15. Male subject and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration. Two acceptable methods of birth control thus include the following:

    * Condom (barrier method of contraception); AND

    One of the following is required:
    * Established use of oral, or injected or implanted hormonal method of contraception by the female partner;
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner;
    * Additional barrier method: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository by the female partner;
    * Tubal ligation in the female partner;
    * Vasectomy or other procedure resulting in infertility (e.g., bilateral orchiectomy), for more than 6 months
16. Subjects must have normal organ and marrow function as defined below:

    * absolute neutrophil count >1,500/µL
    * platelets >100,000/µL
    * total bilirubin <2.5 X institutional upper limit of normal
    * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
    * Creatinine ≤ 2.0 OR creatinine clearance >30 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.

Exclusion Criteria:

1. Definite evidence of metastatic prostate cancer, in the opinion of the treating physician. Pelvic and retroperitoneal lymph nodes < 2.0 cm in short axis are allowed.
2. Subjects who have had treatments with GnRH agonists/antagonists and/or anti-androgens within 1 year of randomization.
3. Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA values (e.g., saw palmetto) or systemic corticosteroids for prostate cancer within 4 weeks of day 29 visit (start of Enzalutamide and ADT).
4. Subjects who have had radiotherapy within 12 weeks prior to entering the study or those who have not recovered from adverse events due to agents or therapies administered for treatment of prostate cancer more than 4 weeks earlier (except urinary, rectal, and sexual side effects related to prostatectomy or radiotherapy are permitted)
5. Subjects who have had any surgical procedure (i.e. TURP, etc.) within 4 weeks prior to entering the study.
6. Subjects who are receiving any other investigational agents.
7. Significant cardiovascular disease, including:

   * Symptomatic left ventricular dysfunction or known baseline left ventricular ejection fraction (LVEF) by multigated acquisition scan (MUGA) or echocardiogram (ECHO) of < lower limit of institutional normal (LLN). "Symptomatic" is defined as New York Heart Association (NYHA) Class II or greater. Note: MUGA and ECHCO do NOT need to be measured to establish eligibility for this study.
   * Uncontrolled hypertension (in the opinion of the treating provider).
   * Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug.
   * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) within 12 months of first dose of study drug.
   * Uncontrolled cardiac arrhythmias.
   * Coronary or peripheral artery bypass graft within 6 months of first dose of study drug.
   * History of CVA, TIA, or rest claudication within 6 months of first dose of study drug.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements (in the opinion of the treating provider).
9. Subjects with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs the ability to swallow and retain enzalutamide are excluded.
10. History of another invasive cancer within 5 years of randomization with the exceptions of (a) non-melanoma skin cancers and (b) American Joint Committee on Cancer (AJCC) Stage 0 or 1 cancers that have a remote probability of recurrence, in the opinion of the treating physician, in consultation with the principal investigator.
11. Known or suspected brain metastasis or leptomeningeal disease.
12. History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma) at any time in the past. Also, history of loss of consciousness or transient ischemic attack within 12 months of the Day 1 visit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Harrison MR, Davis PG, Khouri MG, Bartlett DB, Gupta RT, Armstrong AJ, McNamara MA, Zhang T, Anand M, Onyenwoke K, Edwardson S, Craig D, Michalski M, Wu Y, Oyekunle T, Coyne B, Coburn A, Jones LW, George DJ. A randomized controlled trial comparing changes in fitness with or without supervised exercise in patients initiated on enzalutamide and androgen deprivation therapy for non-metastatic castration-sensitive prostate cancer (EXTEND). Prostate Cancer Prostatic Dis. 2022 Mar;25(1):58-64. doi: 10.1038/s41391-022-00519-4. Epub 2022 Mar 10. PMID 35273377

RESULTS

PARTICIPANT FLOW:
Groups:
- ENZ+ADT+Usual Care: The usual care arm will receive treatment with enzalutamide with androgen deprivation therapy, with no supervised exercise training.
  Enzalutamide
  Androgen deprivation therapy
- ENZ+ADT+Exercise: The ENZ+ADT+Exercise arm will receive treatment with enzalutamide plus androgen deprivation therapy along with supervised exercise training.
  Enzalutamide
  Androgen deprivation therapy
  Supervised exercise training
Period: Overall Study
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.37 (8.31) | 65.66 (8.11) | 65.01 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in VO2peak in Usual Care Versus Exercise Training Arms
Description: Mean change in peak oxygen uptake (VO2peak) from week 1 to week 17 in the usual care and exercise training groups
Time Frame: From week 1 to week 17
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 13 | 13
mL/kg/min | -3.23 (5.02) | -0.92 (2.4)

2. Secondary Outcome: 17-week Change in Functional Capacity as Measured by Chair-stand Test
Description: Mean change in number of seconds to perform the chair-stand test between baseline and week 17. This test measures the time taken to complete 5 repetitions of the sit-to-stand maneuver from a chair without an arm rest at 43 cm in height and 47.5 cm in depth. This test provides an indicator of functional performance of lower body strength; quicker times indicate greater strength
Time Frame: Baseline to 17 weeks
Population: One patient in the usual care arm did not complete the test at week 17
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 12 | 13
seconds | -1.08 (2.29) | -0.78 (1.7)

3. Secondary Outcome: 17-week Change in Upper and Lower Extremity Maximal Muscular Strength
Description: Mean change in upper and lower extremity maximal muscular strength as measured by the voluntary one-repetition max (1-RM) and muscular endurance as measured by 70% of 1-RM between week 17 and baseline
Time Frame: Baseline to 17 weeks
Population: 1 patient out of 13 did not complete the 1-RM at baseline or week 17 in the usual care arm, and another did not complete the 70% 1-RM at week 17 out of 12
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 12 | 13
pounds
  Change in Leg Press 1-RM | 6.67 (83.99) | 107.8 (105.75)
  Change in Leg Press 70% 1-RM | 10 (57.4) | 74.92 (74.05)
  Change in Chest Press 1-RM | 5.08 (24.96) | 24.31 (24.99)
  Change in Chest Press 70% 1-RM | 6.73 (13.93) | 17 (17.32)
  Change in Seated Row 1-RM | 2.25 (20.86) | 14.85 (23.39)
  Change in Seated Row 70% 1-RM | -0.27 (18.29) | 10.46 (16.47)

4. Secondary Outcome: Effects on Serum Glucose
Description: Mean change in fasting serum glucose between week 17 and baseline.
Time Frame: Baseline to 17 weeks
Population: Only 10 in the usual care and 8 in the exercise arm patients had glucose measurements at both baseline and week 17.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 10 | 8
mg/dL | 5.3 (16.22) | -1 (5.55)

5. Secondary Outcome: Change in the Effect on Patient Reported Outcomes (PROs) of Interest Over Time
Description: Mean change in PROs aggregate score between week 17 and baseline. PROs include the FACT-Prostate (FACT-P, range 0 to 104), FACIT-Fatigue (FACIT-F, range 0 to 52), and the Godin Leisure Questionnaire. Higher scores indicate better quality of life.
Time Frame: Baseline to 17 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 13 | 13
score on a scale
  FACIT-Fatigue score | -9.15 (11.25) | -5 (4.88)
  FACT-Prostate Trial Outcome Index | -11.61 (14.39) | -5.38 (9.01)
  Godin Leisure score | 4.67 (26.2) | 9.33 (17.55)

6. Secondary Outcome: Eligibility Rate
Description: Eligibility rate is defined as the number of subjects found to be eligible divided by the number approached for the study. Note that ineligible subjects are not randomized. This is reported as a percent.
Time Frame: 29 months from study initiation
Population: This overall number of participants analyzed reflects the total number of individuals approached for this study.
Measure: Number; unit: percentage of participants
Groups:
- Approached Subjects: The usual care arm will receive treatment with enzalutamide with androgen deprivation therapy, with no supervised exercise training.
  Enzalutamide
  Androgen deprivation therapy
Arm/Group | Approached Subjects
Number analyzed (Participants) | 30
percentage of participants | 87

7. Secondary Outcome: Acceptance Rate
Description: Acceptance rate is defined as the number of patients agreeing to participate divided by total number randomized. This is reported as a percent.
Time Frame: 29 months from study initiation
Measure: Number; unit: percentage of participants
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 13 | 13
percentage of participants | 100 | 100

8. Secondary Outcome: Adherence Rate
Description: Adherence rate is defined as the percentage of days that each patient fulfilled the assigned exercise prescription of the 48 days. The median percentage is reported.
Time Frame: 48 days
Measure: Median (Full Range); unit: percentage of days
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 13 | 13
percentage of days | NA [NA to NA] — Adherence rate does not apply to the usual care arm. | 95.8 [81.2 to 100]

9. Secondary Outcome: Attrition Rate
Description: Attrition rate is defined as the percent of subjects who complete the 16 week exercise training program. This outcome applies only to the exercise arm.
Time Frame: 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 13 | 13
percentage of participants | NA — Attrition rate does not apply to the usual care arm. | 100

10. Secondary Outcome: 17-week Change in Functional Capacity as Measured by Time Up and Go Test
Description: Mean change in number of seconds to complete the timed up and go test between week 17 and baseline. This test requires patients to stand up from a chair with armrests, walk 3m, turn around, return to the chair, and sit down
Time Frame: Baseline to 17 weeks
Population: One patient in the usual care arm did not complete the test at week 17
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 12 | 13
seconds | 0.33 (1.07) | 0.08 (0.95)

11. Secondary Outcome: 17-week Change in Functional Capacity as Measured by Six Minute Walk Test
Description: Mean change in distance covered during the six minute walk test between week 17 and baseline. This test requires patients to cover the longest distance possible in six minutes under the supervision of an exercise physiologist or designee.
Time Frame: Baseline to 17 weeks
Population: Two patients in the usual care arm did not complete the test at both baseline and week 17
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 11 | 13
meters | -32.02 (58.47) | 42 (60.26)

12. Secondary Outcome: 17-week Change in Muscle Cross-sectional Area (CSA)
Description: Mean change in muscle cross sectional area of the dominant quadricep, hamstring, and total mid-thigh between week 17 and baseline. Cross-sectional area was measured using magnetic resonance imaging with a 3.0T-scanner.
Time Frame: Baseline to 17 weeks
Population: Only 10 in the usual care and 8 in the exercise arm patients had cross-sectional area measurements performed at both measurement time points.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 10 | 8
cm^2
  Change in quadricep CSA | -4.84 (4.03) | -4.03 (3.24)
  Change in hamstring CSA | -4.8 (5.32) | -5.09 (4.04)
  Change in total mid-thigh CSA | -9.43 (6.12) | -9.12 (7.01)

13. Secondary Outcome: Effects on Serum Insulin
Description: Mean change in fasting serum insulin between week 17 and baseline.
Time Frame: Baseline to 17 weeks
Population: Only 10 in the usual care and 8 in the exercise arm patients had insulin measurements at both baseline and week 17.
Measure: Mean (Standard Deviation); unit: u[iU]/mL
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 10 | 8
u[iU]/mL | 2.61 (5.06) | 0 (11.05)

14. Secondary Outcome: Effects on Blood Hemoglobin (Hgb)
Description: Mean change in blood hemoglobin (Hgb) A1C between week 17 and baseline.
Time Frame: Baseline to 17 weeks
Population: Only 10 in the usual care and 8 in the exercise arm patients had Hgb measurements at both baseline and week 17.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 10 | 8
percentage of glycated hemoglobin | -0.04 (0.39) | 1.15 (2.81)

15. Secondary Outcome: Effects on Body Composition
Description: Mean change in lean body mass and fat body mass between week 17 and baseline as measured by a DEXA Scan.
Time Frame: Baseline to 17 weeks
Measure: Mean (Standard Deviation); unit: g
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
Number analyzed (Participants) | 13 | 13
g
  Change in lean body mass | -3087.92 (3799.02) | -2094.42 (2407.27)
  Change in fat body mass | 2949.36 (3944.65) | -121.45 (2435.41)

ADVERSE EVENTS:
Time Frame: 37 weeks
Description: Adverse events were collected using Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
Arm/Group | ENZ+ADT+Usual Care | ENZ+ADT+Exercise
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 4/13 | 0/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENZ+ADT+Usual Care (N=13) | ENZ+ADT+Exercise (N=13)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, Specify: RIGHT CORONARY ARTERY STENOSIS (90% OCCULUSION) (Cardiac disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Other, Specify: SURGICAL PROCEDURE FOR INVASIVE ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Surgical and medical procedures - Other, Specify: INGUINAL HERNIA REPAIR, LAPAROSCOPIC (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENZ+ADT+Usual Care (N=13) | ENZ+ADT+Exercise (N=13)
Other, Specify: ABNORMAL ECG (Cardiac disorders) | 1 | 0
Other, Specify: ST DEPRESSION (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Other, Specify: "BURPING" (Gastrointestinal disorders) | 1 | 0
Other, Specify: STOMACH SPASMS (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 11 | 10
Flu like symptoms (General disorders) | 0 | 1
Irritability (General disorders) | 2 | 1
Localized edema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 3 | 2
Other, Specify: SURGICAL WOUND INFECTION FOLLOWING HERNIA REPAIR (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Other, Specify: LEG SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
Other, Specify: MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 1 | 0
Other, Specify: WEAKNESS IN EXTREMITIES (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Cognitive disturbance (Nervous system disorders) | 2 | 2
Concentration impairment (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Hypersomnia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 1
Other, Specify: INTERMITTENT SLEEP DISTURBANCE (Nervous system disorders) | 1 | 0
Other, Specify: VIVID DREAMS (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 6
Libido decreased (Psychiatric disorders) | 0 | 1
Other, Specify: MOODY (Psychiatric disorders) | 1 | 0
Other, Specify: SLEEP DISTURBANCE - NIGHTMARES (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Other, Specify: TROUBLE STARTING STREAM (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 3 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 2 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Gynecomastia (Reproductive system and breast disorders) | 1 | 0
Other, Specify: ERECTION LASTING 14-16 HOURS, NON-PAINFUL. (Reproductive system and breast disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Other, Specify: ABDOMINAL RASH (Skin and subcutaneous tissue disorders) | 0 | 1
Other, Specify: NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0
Other, Specify: PENIS LESION (Skin and subcutaneous tissue disorders) | 0 | 1
Other, Specify: PUBIC HAIR LOSS (R/T RADIATION THERAPY) (Skin and subcutaneous tissue disorders) | 1 | 0
Other, Specify: NUMBNESS IN LOWER RIGHT LIP (Surgical and medical procedures) | 0 | 1
Hot flashes (Vascular disorders) | 12 | 13
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 2 | 0
Other, Specify (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT02256111/Prot_SAP_000.pdf